CLINICAL TRIAL: NCT06774105
Title: The Effects of 6 Weeks of Static Stretching on Blood Glucose and Insulin Sensitivity in People with Type 1 Diabetes
Brief Title: Stretching and Diabetes
Acronym: STREDIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Ewan Thomas, Associate Professor, University of Palermo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 260-2024
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Type 1 diabetes; stretching; insulin sensitivity; insulin requirements; blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CC (No Intervention): The participants continue with their own activities for the study period
- SS (Experimental): The participants undergo a static stretching protocol twice a week for six weeks. The protocol consists in 2 sessions per week, each comprising 8 exercises targeting all major muscle groups: 1) Hamstrings, 2) Knee Extensors, 3) Dorsal muscles, 4) Pectoralis muscles, 5) Elbow Flexors (biceps), 6) Elbow Extensors (triceps), 7) Adductors, and one day 8a) Spine Extensors while the second 8b) Spine Flexors. Each exercise involved 4 sets of 30 seconds of SS and 30 seconds of rest.
  Interventions: Other: Static Stretching

INTERVENTIONS:
Other: Static Stretching — The protocol consisted in 2 sessions per week, each comprising 8 exercises of static stretching targeting all major muscle groups: 1) Hamstrings, 2) Knee Extensors, 3) Dorsal muscles, 4) Pectoralis muscles, 5) Elbow Flexors (biceps), 6) Elbow Extensors (triceps), 7) Adductors, and one day 8a) Spine Extensors while the second 8b) Spine Flexors. Each exercise involved 4 sets of 30 seconds of SS and 30 seconds of rest.
  Arms: SS

SUMMARY:
Diabetes mellitus is a persistent disease characterized by alterations in glucose metabolism due to insufficient insulin production or decreased sensitivity to insulin. Exercise is the most effective non-pharmacological intervention to manage glucose levels and improve insulin sensitivity in people with diabetes. However, little is known regarding the potential effects of stretching. The objective of this study was to understand if six weeks of whole body static stretching could be adopted to manage glycemia and improve insulin sensitivity in a sample of active people with type 1 diabetes.

DETAILED DESCRIPTION:
Diabetes mellitus is a persistent disease characterized by alterations in glucose metabolism due to insufficient insulin production or decreased sensitivity to insulin. The main forms are type 1 (T1D) and type 2 diabetes (T2D). T1D, or juvenile diabetes, represents about 5-10% of cases and is characterized by autoimmune destruction of pancreatic beta cells, which are responsible for insulin production. Managing the disease requires constant monitoring and strict control of blood glucose levels. T1D patients need lifelong external insulin administration to compensate for the lack of internal production.

Physical activity (PA) is one of the most effective non-pharmacological methods to prevent diabetes mellitus and treat cardiometabolic conditions associated with this condition. A multicenter study highlighted that regular PA in patients with T1D improves glycemic control. PA influences glucose levels, offering a means to prevent or avoid the worsening of diabetic complications. Regular PA leads to skeletal muscle adaptations that increase muscle sensitivity to glucose uptake, reducing the need for insulin. Despite the benefits of physical activity on cardiometabolic components and quality of life for patients with T1D, over 50% of these patients do not meet the recommended levels of PA.

Among the most popular forms of PA are aerobic and resistance training (RT). Aerobic training is inversely related to the risk of cardiovascular disease and all-cause mortality in T1D, but this latter type of training, especially of medium-low intensity (for long periods), can lead to hypoglycemia, especially if insulin doses and carbohydrate intake are not adjusted to training needs. In contrast, intense RT, generally causes an increase in blood sugar levels due to the release of catecholamines. On the other hand, the benefits of RT in the management and control of T1D are well known. RT of either moderate or high intensity, can offer multiple benefits to people with T1D which include increased muscle strength, improved lipid profile, decreased insulin dosage, and reduced blood glucose levels. A systematic review and meta-analysis found that RT is associated with a significant reduction in glycated haemoglobin (HbA1c), an indicator of long-term glycemic control, compared to control groups. RT can also improve insulin sensitivity in individuals with T1D and reduce the risk of exercise-induced hypoglycemia following aerobic exercise.

Another type of training that has traditionally been used to improve range of movement (ROM) is stretching. Stretching, compared to other forms of exercise, can be performed in a more static setting, and it may be adopted as a suitable alternative for both rehabilitative environments and specific conditions that prevent autonomous exercise. Recent evidence has shifted from the traditional focus of stretching on improving flexibility to broader systemic effects. In this regard, it has been observed that stretching-based interventions can significantly reduce blood glucose levels and HbA1c, regardless of the type of stretching. The review highlighted that the effects were more evident in patients with T2D. Despite the insights provided by this latter review article, there are no known effects of stretching interventions on glucose management and insulin sensitivity in patients with T1D. Since hypoglycemia is the primary barrier to exercise in this population, event that does not occur in T2D patients, it is crucial to evaluate exercise-specific responses in individuals with T1D. Therefore, our study aims to determine if a 6-week whole body static stretching (SS) intervention can be used as an exercise intervention to manage glycemia and improve insulin sensitivity in a sample of active people with T1D.

Data concerning blood glucose levels (mg/dl), daily CHO consumption and UI/die will be extracted from the continuous glucose monitor of each participant. CGM systems allow people with T1D to monitor in real-time changes in blood glucose. All participants have to be experienced in carbohydrate counting. However, to increase consistency a mobile phone app will be recommended (Yazio for Ios and Android) that extracted the grams of CHO by providing the amount and type of food ingested. UI/die will also be calculated as a sum of basal and bolus insulin units injected per day. The insulin sensitivity index (IS) will then be calculated as the CHO-to-UI/die ratio, which was calculated as the total grams of CHO consumed during one day to the total UI/die.

Participants will be assigned to two groups: a CC and an experimental group. The CC will maintaine their usual exercise routine, while the experimental group will include to their usual exercise routine, during non-training days, a 6-week SS exercise protocol. The protocol will consist in 2 sessions per week, each comprising 8 exercises targeting all major muscle groups: 1) Hamstrings, 2) Knee Extensors, 3) Dorsal muscles, 4) Pectoralis muscles, 5) Elbow Flexors (biceps), 6) Elbow Extensors (triceps), 7) Adductors, and one day 8a) Spine Extensors while the second 8b) Spine Flexors. Each exercise 4 sets of 30 seconds of SS and 30 seconds of rest. Before each session, blood glucose levels will be monitored to ensure stability. In cases participants will show signs of impending hypoglycemia, sessions will be interrupted.

ELIGIBILITY:
Inclusion Criteria:

1. have a diagnosis of type 1 diabetes from at least 1 year
2. exercise regularly 2 to 3 times per week
3. perform exercise activities other than stretching
4. absence of other diabetes-related diseases or comorbidities that prevent them from safely exercising
5. HbA1c level ≤ 7%
6. BMI ≤ 29.9 kg/m²
7. use a CGM reader to monitor glucose levels and daily CHO intake (g) and insulin administration (IU/die).

Exclusion Criteria:

1. have a diagnosis of type 1 diabetes from less than 1 year
2. exercise less or more than 2 to 3 times per week
3. perform stretching exercises during the study period
4. presence of other diabetes-related diseases or comorbidities that prevent them from safely exercising
5. HbA1c level greater than 7%
6. BMI greater than 29.9 kg/m²
7. not using a CGM reader to monitor glucose levels and daily CHO intake (g) and insulin administration (IU/die).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | From enrollment to the end of treatment at 6 weeks

SECONDARY OUTCOMES:
Insulin Requirements | From enrollment to the end of treatment at 6 weeks
Insulin Sensitivity | From enrollment to the end of treatment at 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Palermo, Palermo, IT, Italy

IPD SHARING:
Plan to Share IPD: No
The data will not be publicly available; however, data will be shared upon request with the corresponding author if required.